CLINICAL TRIAL: NCT02592148
Title: Collection of Saliva and Blood Samples From Voluntary Donors to Establish the Occurrence of Selected Vitamins in Saliva and to Investigate Their Concentration Relative to Blood Levels
Brief Title: Occurrence of Selected Vitamins in Saliva and Blood
Acronym: SaliVit
Status: Completed | Type: Observational
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BTS829/14
Record Dates: First submitted 2015-10-26; First posted 2015-10-30 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Divorced State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Health subjects: Male and female

SUMMARY:
There is an interest to assess nutritional status of vitamins in humans in a non-invasive way, i.e. by avoiding taking blood samples. Saliva could potentially be an alternative to blood for this purpose. The suitability of saliva for status determination will be investigated by analysis of (forms of) vitamins A and E, B1, B2, B3, B6 and C in both saliva and blood.

DETAILED DESCRIPTION:
There is an interest to assess nutritional status of vitamins in humans in a non-invasive way, i.e. by avoiding taking blood samples. Saliva could potentially be an alternative to blood for this purpose. However, literature data on vitamins in saliva is scarce. The occurrence is best demonstrated for 25-hydroxy-vitamin D3 where already indications for a correlation to blood levels have been observed in a small scale supplementation study. Occurrence of (forms of) vitamins A and E, B1, B2, B3, B6 and C has been reported but is less well documented. Some information is somewhat ambiguous and for none of these latter vitamins blood levels have been investigated in parallel to saliva.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy males and females
* Age: 20-65 years
* Non-smokers
* No recent or recently (within the last four weeks) started intake of vitamin supplements; long-term intake of supplements on regular base is o.k., but needs to be documented (type of supplement and dosage)
* Subjects willing and able to give written informed consent and to understand, to participate and to comply with the biomedical research project requirements.

Exclusion Criteria:

* Any condition that, in the investigator's opinion would impact volunteer safety and/or a volunteer's ability to complete all study related procedures. (e.g. psychiatric illness, drug addiction, alcoholism, etc.)
* Known infection with human immunodeficiency virus (HIV) or hepatitis.
* Chronic intake of substances affecting blood coagulation (e.g. acetylic acid, anticoagulants, diuretics, thiazides), which in the investigator's opinion would impact volunteer safety
* Allergy or known hypersensitivity against disinfection solutions
* Women: pregnancy, or during lactation
* Currently participating in another study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 50 subjects (females and males, with at least 40% of each gender) generally regarded as healthy in the age of 20 - 65 years.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Identify and quantify selected forms of vitamins in saliva and blood/plasma samples | 1 day
  Selected forms of vitamins: vitamins A (retinol), E (alpha-tocopherol), D (25-hydroxy-vitamin D3), B1 (thiamine), B2 (riboflavine, FAD and FMN), B3 (nicotinic acid and nicotinamide), B6 (pyridoxal and pyridoxamine) and C (ascorbic acid). The measurement of this vitamin concentrations in blood/plasma and saliva will add to our knowledge of the occurrence or absence of these vitamins in saliva, and their concentration levels. Such information is only scarce in literature. Concentrations will be reported in ng/ml or microg/ml for each subject, and as mean for all participants.
  Sampling of saliva, blood and plasma takes place at one time point only. Samples will be measured and reported within 3 month

SECONDARY OUTCOMES:
Determination of the relationship of saliva and blood/plasma concentrations of vitamins A, E, D, B1, B2, B3, B6 and C. | 1 day
  Concentrations measured in saliva and blood/plasma will be correlated to by e.g. linear regression models. The correlation coefficients will be reported. They give an indication on a possible positive relationship of saliva and blood/plasma status of vitamins in humans.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, Dr., Principal Investigator — BioTeSys
Locations (1):
- BioTeSys, Esslingen am Neckar, Germany